CLINICAL TRIAL: NCT05485428
Title: Home-based High-intensity Interval Training for People With Parkinson's: The HIIT-Home4Parkinson's Randomised Controlled Feasibility Study
Brief Title: The HIIT-Home4Parkinson's Study
Acronym: HH4P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Plymouth (Other)
Responsible Party: Principal Investigator, (Ivan) Conrad Harpham, PhD student, Principal Investigator, University of Plymouth
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UPlymouthCH
Record Dates: First submitted 2022-07-27; First posted 2022-08-03 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Parkinson's Disease
Keywords: HIIT; Exercise; Neurodegenerative; Physical; High-intensity; Interval; Home-based; Training
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Randomised controlled feasibility study with mechanistic, physiological and clinical sub components
Who Masked: Outcomes Assessor
Masking Description: Assessor blinded to group allocation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): High-intensity interval training plus usual care
  Interventions: Other: High-intensity interval training
- Usual care (No Intervention): Usual care / treatment. Usual physical activity.

INTERVENTIONS:
Other: High-intensity interval training — 12-weeks of high intensity interval exercise, 30 minutes thrice weekly
  Arms: Exercise

SUMMARY:
This project aims to investigate the practicality and utility of home-based high-intensity interval training (HIIT) by undertaking a previously developed, novel home-based HIIT intervention for people with Parkinson's (PwP).

DETAILED DESCRIPTION:
This is a randomised controlled feasibility study with mechanistic, physiological and clinical sub components.

Participants will be undertaking a 12-week home-based high-intensity interval training intervention. The programme is a feasibility study, previously co-created by people with Parkinson's and clinicians within an iterative planning process of focus groups and exercise testing.

Following recruitment, participants will undertake initial baseline assessments. These will involve collection of anthropometric measurements and general lifestyle and Parkinson's related information, followed by pre-intervention mechanistic, physiological and clinical outcome measures. Participants will then be randomised to the HIIT intervention, or usual care control group.

Both groups will then undertake 7 days pre-intervention physical activity monitoring following accelerometer instruction, as a baseline measure of habitual physical activity (an important confounding variable).

Following an initial home visit, participants will then undertake a 12-week high-intensity interval training programme in the home setting, with supplied exercise equipment including music and exercise prompts, and remote support and online resources. Participants will complete a 32 minute training session 3 times per week, with at least one day of rest between sessions. Participants will be loaned heart rate monitoring devices, which will remotely record heart rate per exercise session. During week 7 of the intervention, participants will be asked to repeat 7 days of accelerometer wearing to compare habitual physical activity. Participants will record feasibility and safety aspects such as HIIT participation / adverse effects and events / exercise adaptations in diaries during the course of the intervention.

Participants will then undergo post-intervention outcome measures. Participants will also be asked to be involved in a 45-minute post intervention focus group as part of a process evaluation. Depending on numbers, it is likely that there will be 2 of these parallel groups.

ELIGIBILITY:
Inclusion criteria:

* Diagnosed with Parkinson's disease
* Aged 18 years or older (No upper limit)
* Hoehn and Yahr stages 1-3 (Mild to moderate disease severity)
* Capacity to consent under the Mental Capacity Act 2005, and able to follow an exercise programme
* Based at home with enough space to perform an exercise programme
* Willing and able to travel to intervention assessments
* Access to a computer, Smart Phone, or tablet and to the internet.

Exclusion criteria:

* Other concurrent neurological condition
* Co-morbidities that would prevent / be exacerbated by high-intensity exercise such as forms of cardiovascular disease
* Advised to not participate following medical consultation
* Participation in a contemporaneous interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Programme completion | Through study completion, an average of 12 weeks
  Number of weeks of exercise programme completed, self administered
Programme adherence | Through study completion, an average of 12 weeks
  Number of exercise sessions completed in full, self administered
Change from baseline brain derived neurotrophic factor (BDNF) | 1 week before first exercise session and 1 day after last session.
  Blood sample: Brain-derived neurotrophic factor (pg/ml)
Change from baseline Relative VO2max | 1 week before first exercise session and 1 day after last session.
  Maximal oxygen uptake (ml/min/kg) incremental exercise test

SECONDARY OUTCOMES:
Adverse effects and events | Through study completion, an average of 12 weeks
  Adverse effects and events related to exercise sessions, self administered
Change from baseline 30 second sit to stand test | 1 week before first exercise session and 1 day after last session.
  Number of times standing in 30 seconds
Oxford Participation Activities Questionnaire | 1 week before first exercise session and 1 day after last session
  Participant administered lifestyle questionnaire
Change from baseline Movement Disorder Society Unified Parkinson's Disease Rating Scale part 3 | 1 week before first exercise session and 1 day after last session.
  Motor examination, minimum score 0, maximum score 76, higher scores indicate increased disease severity
Exercise intensity | Through study completion, an average of 12 weeks
  Achieved exercise intensity (% of maximum heart rate), self administered

OTHER OUTCOMES:
Total weekly habitual physical activity | 1 week prior to start of exercise programme after baseline assessments
  Weekly physical activity (minutes) measured with accelerometer, self administered
Total weekly habitual physical activity | During week 7 of the exercise programme
  Weekly physical activity (minutes) measured with accelerometer, self administered
Maximum heart rate | 1 week before first exercise session
  Beats per minute, to be measured during VO2max assessment
Height | 1 week before first exercise session
  Height (centimetres) with stadiometer
Weight | 1 week before first exercise session
  Weight (kilograms) with calibrated digital scales
Lifestyle data questionnaire | 1 week before first exercise session
  10-item basic lifestyle data bespoke questionnaire
Health screening questionnaire | 1 week before first exercise session at baseline assessments
  Screening for health issues that may prevent participation

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Plymouth NHS Trust, Plymouth, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: De-identified data will be available for a period of 10 years in line with University of Plymouth policy
Access Criteria: On request

REFERENCES:
- [Derived] Harpham C, Gunn H, Marsden J, Bescos-Garcia R, Murgatroyd C, Connolly L. Home-Based High-Intensity Interval Training for People With Parkinson's: A Randomized, Controlled, Feasibility Trial. Health Sci Rep. 2025 Jul 14;8(7):e71024. doi: 10.1002/hsr2.71024. eCollection 2025 Jul. PMID 40661734